CLINICAL TRIAL: NCT03720665
Title: Cortical Excitability Changes on the Sensorimotor Cortex Induced by Caffeine Consumption: A TMS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Walter Paulus, Prof. Dr., University Medical Center Goettingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UMCGoettingen
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Cortical Excitability; Brain Stimulation

STUDY DESIGN:
Intervention Model Description: 15 participants are assigned to caffeine group and another 15 are assigned to placebo group. Then, the participants who were initially in the caffeine group now be in placebo group and those who were in the placebo group were assigned to caffeine group. Finally, all participants received both placebo and caffeine
Who Masked: Participant, Investigator
Masking Description: A statistician prepares a randomization list. Only pharmacist knows the medication type (caffeine or placebo) and the type of electrical stimulation. An investigator is blinded to the type of electrical stimulation and medication. In addition, all participants are naive to electrical stimulation and does not know type of medications that they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine group (Active Comparator): * 200mg caffeine tablet
  * transcranial alternating current stimulation (140 Hz tACS) at 1 mA
  * transcranial alternating current stimulation (140 Hz tACS) at 0.4 mA
  * transcranial alternating current stimulation (140 Hz tACS) sham
  * paired associative stimulation (PAS 25)
  Interventions: Combination Product: Caffeine_TMS
- Placebo group (Placebo Comparator): * Non-active tablet
  * transcranial alternating current stimulation (140 Hz tACS) at 1 mA
  * transcranial alternating current stimulation (140 Hz tACS) at 0.4 mA
  * transcranial alternating current stimulation (140 Hz tACS) sham
  * paired associative stimulation (PAS 25)
  Interventions: Combination Product: Caffeine_TMS

INTERVENTIONS:
Combination Product: Caffeine_TMS — Caffeine group: participants will receive a caffeine tablet and all electrical stimulations in a random order [transcranial electrical stimulation (tACS 140 Hz at 1 mA, 0.4 mA, sham) and paired associative stimulation (PAS 25)] Placebo tablet: participants will receive a placebo tablet and all electrical stimulations in a random order [transcranial electrical stimulation (tACS 140 Hz at 1 mA, 0.4 mA, sham) and paired associative stimulation (PAS 25)]

SUMMARY:
Caffeine is a widely used psychostimulant drug and acts as a competitive antagonist at adenosine receptors. Its effect is on neurons and glial cells of all brain areas. Chronic consumption of caffeine leads to tolerance which might be associated with an increased number of binding sites in the brain. In deep brain stimulation (DBS), the production of adenosine following the release of adenosine triphosphate (ATP) explains the reduction of in tremor. Binding of adenosine to adenosine A1 receptor suppresses excitatory transmission in the thalamus and thus reduces both tremor-and DBS-induced side effects. Also, the effect of adenosine was attenuated following the administration of the 8-Cyclopentyl-1,3-dipropylxanthine (DPCPX) adenosine A1 receptor antagonist. Therefore, the presence of a receptor antagonist such as caffeine was suggested to reduce the effectiveness of deep brain stimulation (DBS) in treating tremor and other movement disorders.

In light with this finding, we anticipate that the antagonistic effect of caffeine is a culprit to the reduction of effectiveness of any stimulation protocol in non-invasive stimulation (NIBS). In particular the excitatory effects of a NIBS protocol can tentatively be blocked in the presence of caffeine.

In this study, the effects of caffeine consumption on cortical excitability at the sensorimotor cortex shall be examined on focal and non-focal plasticity. Focal plasticity will be induced by paired associated stimulation (PAS) and global cortical plasticity from transcranial alternating current (tACS) stimulation. In case of tACS stimulation, 1) an excitatory protocol (tACS, 140 Hz, 1 mA) and 2) an inhibitory protocol (tACS, 140 Hz, 0.4 mA) with the active electrode over M1 and the return electrode over the orbitofrontal cortex will be used. Changes in cortical excitability are assessed using transcranial magnetic stimulation (TMS) recordings.

Research goals are to examine the effects of caffeine consumption on sensorimotor cortical excitability and stimulation induced plasticity. In addition, this study explores further factors which usually contribute to variability in cortical excitability studies. The results are expected to give a useful recommendation for researchers to reduce confounding factors and hereby improves repeatability.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy participants between the ages of 18-45.
* Right-handed (Oldfield 1971).
* Free willing participation and written, informed consent of all subjects obtained prior to the start of the study.
* Participant who willingly stop consuming caffeinated drinks at least three days before the experiment is performed
* Participant's weight is above 60 kg

Exclusion Criteria:

* Age < 18 or > 45 years old;
* Left hand dominant;
* Evidence of a chronic disease or residuals of a disorder of the nervous system in the history, in particular
* stroke
* History of epileptic seizures;
* Pacemaker or deep brain stimulation;
* Metal implants in the head region (metal used in the head region, for example, clips after the operation of an intracerebral aneurysm (vessel sacking in the region of the brain vessels), implantation of an artificial auditory canal);
* Cerebral trauma with loss of consciousness in prehistory;
* Existence of a serious internal (internal organs) or psychiatric (mental illness)
* Alcohol, medication or drug addiction;
* Receptive or global aphasia (disturbance of speech comprehension or additionally of speech);
* Participation in another scientific or clinical study within the last 4 weeks;
* Pregnancy
* Still period
* Participant who is unable to tolerate with caffeine or coffee products
* Participant who has abnormal heart activity from an electrocardiography (ECG) finding
* Weight is less than 60 kg

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Cortical excitabiliy changes induced by caffeine consumption | Baseline (pre-measurement), immediately after intervention, 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes, 60 minutes
  Amplitude of motor evoked potential change (MEP)

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor (BDNF) gene polymorphisms on cortical plasticity | 3-6 months
  Valine (Val) and Methionine (Met) alleles (i.e. Val66Met; Val66Val; Met66Met; Met66Val)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Paulus, Prof. Dr, Principal Investigator — University of Goettingen
Locations (1):
- Prof. Dr. Walter Paulus, Goettigen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Bekar L, Libionka W, Tian GF, Xu Q, Torres A, Wang X, Lovatt D, Williams E, Takano T, Schnermann J, Bakos R, Nedergaard M. Adenosine is crucial for deep brain stimulation-mediated attenuation of tremor. Nat Med. 2008 Jan;14(1):75-80. doi: 10.1038/nm1693. Epub 2007 Dec 23. PMID 18157140
- [Background] Cappelletti S, Piacentino D, Sani G, Aromatario M. Caffeine: cognitive and physical performance enhancer or psychoactive drug? Curr Neuropharmacol. 2015 Jan;13(1):71-88. doi: 10.2174/1570159X13666141210215655. PMID 26074744
- [Background] Cappelletti S, Piacentino D, Fineschi V, Frati P, Cipolloni L, Aromatario M. Caffeine-Related Deaths: Manner of Deaths and Categories at Risk. Nutrients. 2018 May 14;10(5):611. doi: 10.3390/nu10050611. PMID 29757951
- [Background] Feurra M, Paulus W, Walsh V, Kanai R. Frequency specific modulation of human somatosensory cortex. Front Psychol. 2011 Feb 2;2:13. doi: 10.3389/fpsyg.2011.00013. eCollection 2011. PMID 21713181
- [Background] Higdon JV, Frei B. Coffee and health: a review of recent human research. Crit Rev Food Sci Nutr. 2006;46(2):101-23. doi: 10.1080/10408390500400009. PMID 16507475
- [Background] Marquez-Ruiz J, Leal-Campanario R, Sanchez-Campusano R, Molaee-Ardekani B, Wendling F, Miranda PC, Ruffini G, Gruart A, Delgado-Garcia JM. Transcranial direct-current stimulation modulates synaptic mechanisms involved in associative learning in behaving rabbits. Proc Natl Acad Sci U S A. 2012 Apr 24;109(17):6710-5. doi: 10.1073/pnas.1121147109. Epub 2012 Apr 9. PMID 22493252
- [Background] Moliadze V, Antal A, Paulus W. Boosting brain excitability by transcranial high frequency stimulation in the ripple range. J Physiol. 2010 Dec 15;588(Pt 24):4891-904. doi: 10.1113/jphysiol.2010.196998. PMID 20962008
- [Background] Moliadze V, Antal A, Paulus W. Electrode-distance dependent after-effects of transcranial direct and random noise stimulation with extracephalic reference electrodes. Clin Neurophysiol. 2010 Dec;121(12):2165-71. doi: 10.1016/j.clinph.2010.04.033. Epub 2010 Jun 15. PMID 20554472
- [Background] Moliadze V, Atalay D, Antal A, Paulus W. Close to threshold transcranial electrical stimulation preferentially activates inhibitory networks before switching to excitation with higher intensities. Brain Stimul. 2012 Oct;5(4):505-11. doi: 10.1016/j.brs.2011.11.004. Epub 2012 Feb 22. PMID 22445135
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259
- [Background] Stefan K, Kunesch E, Cohen LG, Benecke R, Classen J. Induction of plasticity in the human motor cortex by paired associative stimulation. Brain. 2000 Mar;123 Pt 3:572-84. doi: 10.1093/brain/123.3.572. PMID 10686179
- [Background] Stefan K, Kunesch E, Benecke R, Cohen LG, Classen J. Mechanisms of enhancement of human motor cortex excitability induced by interventional paired associative stimulation. J Physiol. 2002 Sep 1;543(Pt 2):699-708. doi: 10.1113/jphysiol.2002.023317. PMID 12205201
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- [Derived] Zulkifly MFM, Merkohitaj O, Brockmoller J, Paulus W. Confounding effects of caffeine on neuroplasticity induced by transcranial alternating current stimulation and paired associative stimulation. Clin Neurophysiol. 2021 Jun;132(6):1367-1379. doi: 10.1016/j.clinph.2021.01.024. Epub 2021 Mar 10. PMID 33762129
- [Derived] Zulkifly MFM, Merkohitaj O, Paulus W, Brockmoller J. The roles of caffeine and corticosteroids in modulating cortical excitability after paired associative stimulation (PAS) and transcranial alternating current stimulation (tACS) in caffeine-naive and caffeine-adapted subjects. Psychoneuroendocrinology. 2021 May;127:105201. doi: 10.1016/j.psyneuen.2021.105201. Epub 2021 Mar 15. PMID 33740589